CLINICAL TRIAL: NCT04245098
Title: Carpal Tunnel Syndrome and Amyloidosis
Acronym: AMICAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Maria del Carmen Navarro-Saez, Principal Investigator, Corporacion Parc Tauli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CSPT_AMICAR1
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Amyloidosis; Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; amyloidosis
MeSH Terms: conditions — Amyloidosis; Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amyloid (Experimental): Biopsy
  Interventions: Procedure: Carpal tunnel syndrome surgery

INTERVENTIONS:
Procedure: Carpal tunnel syndrome surgery — Biopsy

SUMMARY:
Carpal tunnel syndrome has been suggested to be an early sign of amyloidosi. The investigators will evaluate tissue samples obtained from patients undergoing carpal tunnel release surgery for amyloid.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) can be caused by the deposition and accumulation of misfolded proteins called amyloid and is often an early manifestation of systemic amyloidosis.

Patients with cardiac amyloidosis often have carpal tunnel syndrome that precedes cardiac manifestations by several years, and many patients will have undergone surgery for idiopathic carpal tunnel syndrome since the protein also deposits in the transversal carpal ligament of the hand.

The investigators sought to identify the prevalence and type of amyloid deposits in patients undergoing carpal tunnel surgery and evaluate for cardiac involvement

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing carpal tunnel syndrome surgery

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-01-08 (Estimated); Study Completion 2023-01-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with amyloid deposits in patients undergoing carpal tunnel surgery | 2 years
  Prevalence of amyloid deposits in biopsy in patients undergoing carpal tunnel syndrome surgery

SECONDARY OUTCOMES:
Number of participants with cardiac involvement in echocardiogram | 2 years
  Cardiac involment in echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Del Carmen Navarro-Saez, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No